CLINICAL TRIAL: NCT00405587
Title: A Study to Assess Safety, Pharmacokinetics, and Pharmacodynamics of PLX4032 in Patients With Solid Tumors
Brief Title: Safety Study of PLX4032 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plexxikon (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX06-02
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2016-10

CONDITIONS: Malignant Melanoma; Colorectal Carcinoma
MeSH Terms: conditions — Melanoma; Colorectal Neoplasms | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLX4032 (Experimental): Open-label, sequential dose escalation
  Interventions: Drug: PLX4032

INTERVENTIONS:
Drug: PLX4032 — Oral capsules administered BID

SUMMARY:
The primary objective of this FIH study is to assess the safety and pharmacokinetics of PLX4032 in patients with solid tumors. The secondary objective is to assess the pharmacodynamic activity in paired biopsy specimens obtained from patients with malignant melanoma who have the V600E BRAF oncogenic mutation.

DETAILED DESCRIPTION:
Activating mutations of the BRAF gene have been observed in a variety of cancers, including 55-68% of malignant melanomas. In general, oncogenic mutations of BRAF correlate with a poor outcome. PLX4032 is a compound that selectively inhibits oncogenic B-Raf kinase.

Two extension cohorts of patients with confirmed V600E mutations will be recruited, consisting of advanced melanoma and metastatic colorectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumors confirmed histologically whose tumors are refractory to standard therapy, or for whom standard or curative therapy does not exist
* Patients from whom paired melanoma biopsies are planned must have a V600E+ BRAF mutation confirmed prior to the administration of PLX4032
* Previous chemotherapy, immunotherapy, or radiation therapy must have been completed at least 2 weeks prior to starting PLX4032 therapy, and all associated toxicity must be resolved prior to administration of PLX4032
* Patients in the Extension cohorts (melanoma or adenocarcinoma of the colon or rectum) must have both a V600E+ BRAF mutation and measurable disease (by RECIST V 1.0 criteria) prior to the administration of PLX4032. All patients enrolled must provide archival or fresh melanoma tumor biopsy for confirmation of V600E+ BRAF mutation status by TaqMan assay
* ECOG performance status 0 or 1
* Life expectancy ≥ 3 months
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Brain metastases that are progressing or have been documented to be stable for less than 3 months, or for which systemic corticosteroids are required
* Investigational drug use within 28 days of the first dose of PLX4032
* Uncontrolled intercurrent illness
* Refractory nausea and vomiting, malabsorption, or significant bowel resection that would preclude adequate absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-11; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hsu, MD, Study Director — Plexxikon
Locations (7):
- United States (5):
  - University of California Los Angeles, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria

REFERENCES:
- [Result] Flaherty KT, Puzanov I, Kim KB, Ribas A, McArthur GA, Sosman JA, O'Dwyer PJ, Lee RJ, Grippo JF, Nolop K, Chapman PB. Inhibition of mutated, activated BRAF in metastatic melanoma. N Engl J Med. 2010 Aug 26;363(9):809-19. doi: 10.1056/NEJMoa1002011. PMID 20818844
- [Derived] Kopetz S, Desai J, Chan E, Hecht JR, O'Dwyer PJ, Maru D, Morris V, Janku F, Dasari A, Chung W, Issa JP, Gibbs P, James B, Powis G, Nolop KB, Bhattacharya S, Saltz L. Phase II Pilot Study of Vemurafenib in Patients With Metastatic BRAF-Mutated Colorectal Cancer. J Clin Oncol. 2015 Dec 1;33(34):4032-8. doi: 10.1200/JCO.2015.63.2497. Epub 2015 Oct 12. PMID 26460303
- [Derived] Puzanov I, Amaravadi RK, McArthur GA, Flaherty KT, Chapman PB, Sosman JA, Ribas A, Shackleton M, Hwu P, Chmielowski B, Nolop KB, Lin PS, Kim KB. Long-term outcome in BRAF(V600E) melanoma patients treated with vemurafenib: Patterns of disease progression and clinical management of limited progression. Eur J Cancer. 2015 Jul;51(11):1435-43. doi: 10.1016/j.ejca.2015.04.010. Epub 2015 May 13. PMID 25980594
- [Derived] Su F, Viros A, Milagre C, Trunzer K, Bollag G, Spleiss O, Reis-Filho JS, Kong X, Koya RC, Flaherty KT, Chapman PB, Kim MJ, Hayward R, Martin M, Yang H, Wang Q, Hilton H, Hang JS, Noe J, Lambros M, Geyer F, Dhomen N, Niculescu-Duvaz I, Zambon A, Niculescu-Duvaz D, Preece N, Robert L, Otte NJ, Mok S, Kee D, Ma Y, Zhang C, Habets G, Burton EA, Wong B, Nguyen H, Kockx M, Andries L, Lestini B, Nolop KB, Lee RJ, Joe AK, Troy JL, Gonzalez R, Hutson TE, Puzanov I, Chmielowski B, Springer CJ, McArthur GA, Sosman JA, Lo RS, Ribas A, Marais R. RAS mutations in cutaneous squamous-cell carcinomas in patients treated with BRAF inhibitors. N Engl J Med. 2012 Jan 19;366(3):207-15. doi: 10.1056/NEJMoa1105358. PMID 22256804

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment to "Dose Escalation: Original Formulation" was halted based on bioavailability results and the drug was reformulated as microprecipitated bulk powder (MBP) and then the enrollment was resumed in "Dose Escalation: MBP Formulation" arm
Groups:
- Dose Escalation: Original Formulation: Cohorts of 3 to 6 participants received RO5185426 capsules in original (crystalline) formulation at a starting dose of 200 mg BID for 4 weeks. After Day 15 pharmacokinetic assessment and adequate safety and tolerability was shown, next cohort of 3 to 6 participants received 50 % to 100% increased dose of RO5185426 original formulation for 4 weeks. Dose escalation was continued up to 1600 mg BID dose level.
- Dose Escalation: MBP Formulation: Cohorts of 3 to 6 participants received RO5185426 capsules/tablets in MBP formulation at a starting dose of 160 mg BID for 4 weeks. After Day 15 pharmacokinetic assessment and adequate safety and tolerability was shown, next cohort of 3 to 6 participants received 50 % to 100% increased dose of RO5185426 MBP formulation for 4 weeks. Dose escalation was continued up to unacceptable toxicity or disease progression occurred.
- Extension: BRAFV600E- Positive Melanoma: Participants with melanoma tumors that carried the V600E mutation of the v-raf murine sarcoma viral oncogene homologue B1 (BRAF) received RO5185426 capsules/tablets in MBP formulation at a dose of 960 mg BID until disease progression, death, or withdrawal from the study.
- Extension: BRAFV600E- Positive CRC: Participants with CRC that carried the V600E mutation of BRAF received RO5185426 capsules/tablets in MBP formulation at a dose of 960 mg BID until disease progression, death, or withdrawal from the study.
Period: Overall Study
Arm/Group | Dose Escalation: Original Formulation | Dose Escalation: MBP Formulation | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Started | 26 | 30 | 32 | 21
Completed | 0 | 2 | 10 | 1
Not Completed | 26 | 28 | 22 | 20
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Disease Progression | 22 | 23 | 21 | 17
Not completed — Physician Decision | 3 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Radiation induced necrosis | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Participant not dosed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All enrolled participants whether or not they fulfilled the eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Original Formulation | Dose Escalation: MBP Formulation | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC | Total
Number analyzed (Participants) | 26 | 30 | 32 | 21 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (13.75) | 58.0 (14.77) | 50.4 (13.54) | 63.6 (14.86) | 58.6 (15.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 14 | 10 | 46
  Male | 15 | 19 | 18 | 11 | 63

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of RO5185426 on Day 1 - Dose Escalation: Original Formulation
Description: AUC (0-8 hour) was defined as the area under the plasma concentration-time curve from time equals zero (0) to 8 hours post-dose. AUC (0-24 hour) was defined as the area under the plasma concentration-time curve from time equals 0 to 24 hours post-dose. AUC (0-8 hour) and AUC (0-24 hour) were computed using the linear trapezoidal rule.
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: Pharmacokinetic (PK) Population: Participants who received all RO5185426 doses without dose reduction up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome; n=participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Groups:
- Dose Escalation: Original Formulation - 200 mg: Participants received RO5185426 capsules in original (crystalline) formulation at a dose of 200 mg BID for 4 weeks.
- Dose Escalation: Original Formulation - 400 mg: Participants received RO5185426 capsules in original (crystalline) formulation at a dose of 400 mg BID for 4 weeks.
- Dose Escalation: Original Formulation - 800 mg: Participants received RO5185426 capsules in original (crystalline) formulation at a dose of 800 mg BID for 4 weeks.
- Dose Escalation: Original Formulation - 1600 mg: Participants received RO5185426 capsules in original (crystalline) formulation at a dose of 1600 mg BID for 4 weeks.
Arm/Group | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 4 | 4 | 4
ug*hr/mL
  AUC (0-8 hour) (n= 6, 4, 4, 4) | 2.02 (1.03) | 3.28 (1.66) | 4.47 (0.61) | 4.23 (2.0)
  AUC (0-24 hour) (n= 6, 4, 4, 4) | 8.43 (4.84) | 14.86 (7.89) | 21.66 (10.59) | 22.34 (10.59)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of RO5185426 on Day 15 - Dose Escalation: Original Formulation
Description: AUC (0-8 hour) was defined as the area under the plasma concentration-time curve from time equals 0 to 8 hours post-dose. AUC (0-24 hour) was defined as the area under the plasma concentration-time curve from time equals 0 to 24 hours post-dose. AUC (0-8 hour) and AUC (0-24 hour) were computed using the linear trapezoidal rule.
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: PK Population: Participants who received all RO5185426 doses without dose reduction up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome; n=participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Groups:
- Dose Escalation Original Formulation - 200 mg: Participants received RO5185426 capsules in original (crystalline) formulation at a dose of 200 mg BID for 4 weeks.
Arm/Group | Dose Escalation Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 3 | 3 | 4
ug*hr/mL
  AUC (0-8 hour) (n=6, 3, 3, 4) | 9.37 (6.18) | 30.90 (11.44) | 30.58 (7.08) | 33.89 (17.24)
  AUC (0-24 hour) (n= 2, 2, 3, 4) | 46.28 (10.47) | 105.10 (65.41) | 91.01 (26.86) | 101.13 (48.40)

3. Primary Outcome: Peak Concentration (Cmax) of RO5185426 on Day 1 - Dose Escalation: Original Formulation
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8 hours post-morning dose on Day 1, pre-morning dose on Day 2 and Day 8
Population: PK Population: Participants who received all RO5185426 doses without dose reduction up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 4 | 4 | 3
Micrograms per milliliter | 0.37 (0.2) | 0.58 (0.27) | 0.85 (0.06) | 0.73 (0.38)

4. Primary Outcome: Peak Concentration (Cmax) of RO5185426 on Day 15 - Dose Escalation: Original Formulation
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8 hours post-morning dose on Day 15, pre-morning dose on Day 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 3 | 3 | 4
Micrograms per milliliter | 1.34 (0.81) | 4.57 (2.07) | 5.41 (2.26) | 5.34 (3.04)

5. Primary Outcome: Time to Peak Concentration (Tmax) of RO5185426 on Day 1 - Dose Escalation: Original Formulation
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1, pre-morning dose on Day 2 and Day 8
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 4 | 4 | 3
hours | 9.98 [4 to 10] | 4 [4 to 4.25] | 3.01 [2 to 8.08] | 4 [2 to 4]

6. Primary Outcome: Time to Peak Concentration (Tmax) of RO5185426 on Day 15 - Dose Escalation: Original Formulation
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 15, pre-morning dose on Day 16
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 3 | 3 | 4
hours | 0.02 [0 to 2] | 0.5 [0 to 10] | 0 [0 to 2] | 3 [0 to 10]

7. Primary Outcome: AUC of RO5185426 on Day 1 - Dose Escalation: MBP Formulation
Description: as for outcome 1
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Groups:
- Dose Escalation: MBP Formulation - 160 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 160 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation - 240 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 240 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation - 360 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 360 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation - 720 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 720 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation - 960 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 960 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation - 1120 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 1120 mg BID for 4 weeks.
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 6 | 5
ug*hr/mL | 5.98 (3.31) | 15.85 (1.53) | 14.95 (4.99) | 39.09 (35.82) | 39.48 (19.58) | 44.94 (20.88)

8. Primary Outcome: AUC of RO5185426 on Day 15 - Dose Escalation: MBP Formulation
Description: as for outcome 1
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
mcg*hr/mL
  AUC (0-8 hour) (n= 4, 4, 4, 4, 3, 4) | 33.91 (19.14) | 71.64 (30.09) | 114.50 (35.33) | 212.28 (123.24) | 229.96 (42.75) | 536.47 (137.18)
  AUC (0-24 hour) (n= 2, 3, 3, 3, 2, 3) | 87.18 (88.78) | 228.97 (81.03) | 373.94 (94.51) | 622.21 (406.89) | 649.29 (200.95) | 1494.27 (367.68)

9. Primary Outcome: Mean RO5185426 Accumulation Ratios - Dose Escalation: MBP Formulation
Description: Accumulation ratio is the ratio of AUC (0-8 hour) on Day 15 / AUC (0-8 hour) on Day 1.
Time Frame: Day 1 and Day 15: pre-morning dose and at 0.5, 1, 2, 4, and 8 hours post-morning dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 3 | 3
ratio | 4.75 (3.14) | 4.47 (1.57) | 8.66 (5.37) | 8.89 (6.03) | 10.11 (3.09) | 13.86 (4.68)

10. Primary Outcome: Mean RO5185426 Accumulation Ratios - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- Positive CRC
Description: Accumulation ratio is the ratio of AUC (0-8 hour) on Day 15 / AUC (0-8 hour) on Day 1.
Time Frame: Day 1 and Day 15: pre-morning dose and at 0.5, 1, 2, 4, and 8 hours post-morning dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 13 | 13
ratio | 11.61 (4.59) | 9.31 (3.90)

11. Primary Outcome: Cmax of RO5185426 on Day 1 - Dose Escalation: MBP Formulation
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1, pre-morning dose on Day 2 and Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 6 | 5
micrograms per milliliter | 1.14 (0.48) | 2.93 (0.39) | 2.72 (0.94) | 7.2 (6.06) | 7.12 (3.71) | 7.73 (3.54)

12. Primary Outcome: Cmax of RO5185426 on Day 15 - Dose Escalation: MBP Formulation
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 15, and pre-morning dose on Day 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
micrograms per milliliter | 5.16 (2.72) | 11.64 (4.55) | 17.90 (8.01) | 31.15 (15.56) | 34.10 (5.47) | 84.30 (23.51)

13. Primary Outcome: Tmax of RO5185426 on Day 1 - Dose Escalation: MBP Formulation
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1, pre-morning dose on Day 2 and Day 8
Population: Pharmacokinetic (PK) Population: Participants who received all RO5185426 doses without dose reduction up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 6 | 5
hours | 2 [2 to 4] | 3 [1 to 4] | 3.21 [2 to 4.08] | 6.29 [3.92 to 8] | 3.29 [2.03 to 8.02] | 4.33 [2 to 8]

14. Primary Outcome: Tmax of RO5185426 on Day 15 - Dose Escalation: MBP Formulation
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 15, and pre-morning dose on Day 16
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 960 mg | Dose Escalation: MBP Formulation - 1120 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 3 | 4
hours | 1.5 [0 to 4.05] | 2.0 [0 to 8.0] | 4.10 [2.5 to 8.45] | 4.07 [0 to 24] | 4.33 [1.0 to 8.0] | 0.41 [0 to 2.33]

15. Primary Outcome: AUC of RO5185426 on Day 1 - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- Positive CRC
Description: as for outcome 1
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: Phamacokinetic (PK) Population: Participants who received all RO5185426 doses without dose reduction up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome; n=participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 29 | 21
mcg*hr/mL
  AUC (0-8 hour) (n= 29, 21) | 31.35 (15.51) | 31.53 (15.1)
  AUC (0-24 hour) (n= 5, 0) | 108.52 (42.36) | NA (NA) — AUC (0-24) was optional in CRC group as steady state kinetics with respect to AUC (0-8) and AUC (0-24) were previously characterized.

16. Primary Outcome: AUC of RO5185426 on Day 15 - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- Positive CRC
Description: as for outcome 2
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 14 | 13
ug*hr/mL
  AUC (0-8 hour) (n= 14, 13 ) | 289.26 (105.88) | 262.42 (101.37)
  AUC (0-24 hour) (n= 9, 11) | 924.65 (317.71) | 752.64 (314.47)

17. Primary Outcome: Cmax of RO5185426 on Day 1 - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- Positive CRC
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1, pre-morning dose on Day 2 and Day 8
Population: Phamacokinetic (PK) Population: Participants who received all RO5185426 doses without dose reduction up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 29 | 21
microgram/milliliter | 5.84 (2.61) | 5.53 (2.27)

18. Primary Outcome: Cmax of RO5185426 on Day 15 - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- Positive CRC
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 15 and pre-morning dose on Day 16
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 14 | 13
microgram/milliliter | 44.31 (16.38) | 38.55 (15.92)

19. Primary Outcome: Tmax of RO5185426 on Day 1 - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- CRC
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1, pre-morning dose on Day 2 and Day 8
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 29 | 21
hours | 4 [1.92 to 8.25] | 4 [2 to 8.5]

20. Primary Outcome: Tmax of RO5185426 on Day 15 - Extension: BRAFV600E- Positive Melanoma and BRAFV600E- CRC
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 15, and pre-morning dose on Day 16
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Extension: BRAFV600E- Positive Melanoma | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 14 | 13
hours | 1.01 [0.0 to 8.0] | 2.0 [0.0 to 8.0]

21. Primary Outcome: Percentage of Participants With a Confirmed and an Unconfirmed Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) According to RECIST Version (v) 1.0 - Extension: BRAFV600E- Positive Melanoma
Description: BOR of confirmed /unconfirmed (total) response was defined as CR or PR recorded from baseline until disease progression/recurrence according to Response Evaluation Criteria In Solid Tumors (RECIST) v 1.0 criteria. For target lesions (TLs), CR was defined as the disappearance of all TLs, and PR was defined as at least a 30 percent (%) decrease in the sum of longest diameters of the TLs, taking as a reference the baseline (BL) sum of longest diameters. For non-target lesions (NTLs), CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. Confirmed responses were those which were confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met. Percentage of participants with best overall response rate was calculated as the (number of participants with CR or PR) divided by (total number of participants in the cohort), and then multiplied by 100. The 95% Cl was determined using the Pearson-Clopper method.
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to data cutoff (up to 337 days)
Population: Modified ITT population: All participants with a measurable disease at BL and completed at least one post-baseline radiographic assessment or discontinued study medication early due to disease progression were considered evaluable for efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 32
percentage of participants
  Confirmed BOR | 56.3 [37.7 to 73.6]
  Unconfirmed BOR | 81.3 [63.6 to 92.8]

22. Primary Outcome: Percentage of Participants With BOR of CR or PR According to RECIST v1.0 - Extension: BRAFV600E- Positive CRC
Description: BOR of CR or PR was recorded from baseline until disease progression/recurrence according to RECIST v 1.0 criteria. For TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the sum of longest diameters of the TLs, taking as a reference the BL sum of longest diameters. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. Confirmed responses were those which were confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met Percentage of participants with best overall response rate was calculated as the (number of participants with CR or PR) divided by (total number of participants in the cohort), and then multiplied by 100. The 95% Cl was determined using the Pearson-Clopper method.
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to data cutoff (up to 337 days)
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Extension: BRAFV600E- Positive CRC
Number analyzed (Participants) | 20
percentage of participants | 5.0 [0.1 to 24.9]

23. Primary Outcome: Percentage of Participants With BOR of CR or PR According to RECIST v1.0 - Dose Escalation: Original Formulation
Description: BOR of CR or PR was recorded from baseline until disease progression/recurrence according to RECIST v 1.0 criteria. For TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the sum of longest diameters of the TLs, taking as a reference the BL sum of longest diameters. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. Percentage of participants with best overall response rate was calculated as the (number of participants with CR or PR) divided by (total number of participants in the cohort), and then multiplied by 100. The 95% Cl was determined using the Pearson-Clopper method.
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to data cutoff (up to 337 days)
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg
Number analyzed (Participants) | 6 | 6 | 10 | 4
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 10.0 [0.3 to 44.5] | 0 [0 to 0]

24. Primary Outcome: Percentage of Participants With BOR of CR or PR According to RECIST v1.0 - Dose Escalation: MBP Formulation
Description: as for outcome 23
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to data cutoff (up to 337 days)
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation: MBP Formulation -160 mg: Participants received RO5185426 hard gelatin capsules at a dose of 160 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation -240 mg: Participants received RO5185426 hard gelatin capsules at a dose of 240 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation -320 mg: Participants received RO5185426 hard gelatin capsules at a dose of 320 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation -360 mg: Participants received RO5185426 hard gelatin capsules at a dose of 360 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation -720 mg: Participants received RO5185426 hard gelatin capsules at a dose of 720 mg BID for 4 weeks.
- Dose Escalation: MBP Formulation -1120 mg: Participants received RO5185426 hard gelatin capsules at a dose of 1120 mg BID for 4 weeks.
Arm/Group | Dose Escalation: MBP Formulation -160 mg | Dose Escalation: MBP Formulation -240 mg | Dose Escalation: MBP Formulation -320 mg | Dose Escalation: MBP Formulation -360 mg | Dose Escalation: MBP Formulation -720 mg | Dose Escalation: MBP Formulation -1120 mg
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 7 | 6
percentage of participants | 0 [0 to 0] | 25.0 [0.6 to 80.6] | 33.3 [0.8 to 90.6] | 40.0 [5.3 to 85.3] | 28.6 [3.7 to 71.0] | 50.0 [11.8 to 88.2]

25. Secondary Outcome: Duration of CR or PR Using RECIST v 1.0 - Extension BRAFV600E- Positive Melanoma
Description: Duration of response for participants with confirmed CR or PR was the period of time measured between the date that the criteria for objective CR or PR (whichever status was recorded first) was met, and the first date that recurrent or PD was objectively documented (or death if before progression). PD was at least a 20% increase in the sum of longest diameters of TLs taking as reference the smallest sum of longest diameters recorded since the baseline measurements, or the appearance of one or more new lesion(s). In the event of no disease progression or documented death prior to study termination, analysis cutoff, or initiation of confounding anticancer therapy, duration of response was censored at the date of the last evaluable tumor assessment.
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to data cutoff (up to 337 days)
Population: Modified ITT population: Participants with confirmed CR or PR with a measurable disease at BL, and completed at least one post-baseline radiographic assessment or discontinued study medication early due to disease progression were considered. Seven participants were censored for analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 18
days | 227 [150 to NA] — The upper limit of the confidence interval was not estimable because of high number of censored participants.

26. Secondary Outcome: Percentage of Participants With Progression-Free Survival (PFS) Using RECIST v 1.0 - Melanoma Extension Cohort
Description: PFS was the period of time measured from the date of initiation of therapy to the date of the appearance of new metastatic lesions, objective tumor progression, or death if before progression. PD was defined according to the RECIST criteria (v 1.0) as increase by at least 20% in the sum of the longest diameters of each TL, taking as a reference the smallest sum of the longest diameters, reported since the start of treatment, or appearance of one or more new lesions. For Non-TLs, PD was defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Month 1, 3, 4, 6, 9, and Last event (350) days
Population: Modified ITT population: All participants with a measurable disease at BL and completed at least one post-baseline radiographic assessment or discontinued study medication early due to disease progression were considered. Eight participants were censored for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 32
percentage of participants
  Month 1 | 96.9
  Month 3 | 87.5
  Month 4 | 75.0
  Month 6 | 59.4
  Month 9 | 43.3
  1 Year | 16.9
  Last Event (350 Days) | 16.9

27. Secondary Outcome: PFS Using RECIST v1.0 - Extension BRAFV600E Positive Melanoma
Description: PFS was the period of time measured from the date of initiation of therapy to the date of the appearance of new metastatic lesions, objective tumor progression, or death if before progression. PD was at least a 20% increase in the sum of longest diameters of TLs taking as reference the smallest sum of longest diameters recorded since the baseline measurements, or the appearance of one or more new lesion(s). For Non-TLs, disease progression was defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-TLs. In the event of no disease progression or documented death prior to study termination, analysis cutoff, or start of confounding anticancer therapy, PFS was censored at the date of the last evaluable tumor assessment.
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to data cutoff (up to 421 days)
Population: as for outcome 26
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 32
days | 233 [149 to 297]

28. Secondary Outcome: Percentage of Participants Who Died - Extension: BRAFV600E- Positive Melanoma
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to 444 days
Population: Modified ITT Population: All participants with a measurable disease at BL and completed at least one post-baseline radiographic assessment or discontinued study medication early due to disease progression were considered.
Measure: Number; unit: percentage of participants
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 32
percentage of participants
  Month 1 | 0
  Month 3 | 3.1
  Month 4 | 6.2
  Month 6 | 12.7
  Month 9 | 29.4
  Month 12 | 43.2

29. Secondary Outcome: Overall Survival (OS) - Extension: BRAFV600E- Positive Melanoma
Description: OS was the period of time measured from the date of initiation of therapy to the date of the death. In the event of no death prior to study termination or analysis data cutoff, OS was censored at the last known date that the patient was alive as documented on the follow-up case report form. If this date was not available, then the last known alive date from the database was used.
Time Frame: Screening, BL, until PD, or end of efficacy follow-up, up to 444 days
Population: Modified ITT Population: All participants with a measurable disease at BL and completed at least one post-baseline radiographic assessment or discontinued study medication early due to disease progression were considered. Twenty participants were censored for analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 32
days | NA [307 to NA] — The median OS was not reached as less than 50% participants had the event of interest.

30. Secondary Outcome: Time to CR or PR Using RECIST v1.0 - Extension: BRAFV600E- Positive Melanoma
Description: Time to CR or PR was defined as the interval between the date of the first treatment to the date of the first documentation of confirmed CR or PR whichever occurred first, and not the date of confirmation at the subsequent tumor assessment. Time to response = Date of first response - initial dose date + 1.
Time Frame: Screening, BL, and up to 168 days
Population: Modified ITT population: Participants with a confirmed CR or PR with a measurable disease at BL and completed at least one post-baseline radiographic assessment or discontinued study medication early due to disease progression were considered.
Measure: Median (Full Range); unit: days
Arm/Group | Extension: BRAFV600E- Positive Melanoma
Number analyzed (Participants) | 18
days | 56.5 [25 to 168]

31. Secondary Outcome: Mean Dose-Normalized Steady-State AUC of RO5185426 80 mg and 120 mg Capsules - Dose Escalation: MBP Formulation and Extension: BRAFV600E- Positive Melanoma
Description: as for outcome 2
Time Frame: Pre-morning dose and at 0.5, 1, 2, 4, and 8, and 24 hours post-morning dose
Population: The analysis was planned only for those participants who received 80 or 120 mg dose of RO5185426 up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome; n=participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Groups:
- Dose Escalation: MBP Formulation - 80 mg Capsule: Participants received RO5185426 capsules in MBP formulation at a dose of 320 mg BID dose escalation/paired biopsy cohort, or 720 mg BID dose escalation/paired biopsy cohort, or 1120 mg BID dose escalation for 4 weeks.
- Dose Escalation: MBP Formulation and Extension: BRAFV600E- Pos: Participants with melanoma tumors that carried the V600E mutation of the v-raf murine sarcoma viral oncogene homologue B1 (BRAF) received RO5185426 capsules in MBP formulation at a dose of 960 mg BID , or 960 mg BID dose escalation
Arm/Group | Dose Escalation: MBP Formulation - 80 mg Capsule | Dose Escalation: MBP Formulation and Extension: BRAFV600E- Pos
Number analyzed (Participants) | 10 | 19
ug*hr/mL
  AUC (0-8hour) (n= 10, 19) | 0.179 (0.081) | 0.197 (0.091)
  AUC (0-24 hour) (n= 7, 9) | 0.524 (0.233) | 0.482 (0.165)

32. Secondary Outcome: Mean Dose-Normalized Steady-State Cmax of RO5185426 80 mg and 120 mg Capsules - Dose Escalation: MBP Formulation and Extension: BRAFV600E- Positive Melanoma
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1 and 15, pre-morning dose on Day 2 and Day 8, and Day 16
Population: PK Population: The analysis was planned only for those participants who received 80 or 120 mg dose of RO5185426 up to and including Day 15 and provided at least PK assessments up to and including 8 to 10 hours after first dose on Day 15. Number of participants analyzed=participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation: MBP Formulation - 80 mg Capsule | Dose Escalation: MBP Formulation and Extension: BRAFV600E- Pos
Number analyzed (Participants) | 10 | 19
ug/mL | 0.028 (0.012) | 0.030 (0.013)

33. Secondary Outcome: Decrease in Tumor Uptake of 18F-fluorodeoxyglucose (FDG)
Description: Tumor uptake of FDG was assessed by means of positron-emission tomography (PET)
Time Frame: BL and Day 15
Reporting Status: Not Posted

34. Secondary Outcome: Cmax of RO5185426 - Food Effect
Time Frame: Pre-morning dose, 0.5, 1, 2, 4, and 8 hour post-morning dose on Day 1 and 15, pre-morning dose on Day 2, Day 8, and Day 16
Reporting Status: Not Posted

35. Secondary Outcome: Tumor Levels of Phosphorylated Extracellular Signal-Regulated Kinapse (ERK), Cyclin D1, and Ki-67
Description: The immunohisto-chemical analyses of the expression of phosphorylated ERK, cyclin D1, and Ki-67 in tumor-biopsy specimens was performed using hematoxylin and eosin staining.
Time Frame: BL and Day 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: For MBP Formulation, one patient not dosed, so only 29 patients are evaluable for safety measures although at the beginning of the study 30 patients started.
Groups:
- Dose Escalation: MBP Formulation - 320 mg: Participants received RO5185426 capsules in MBP formulation at a dose of 320 mg BID for 4 weeks.
- Extension: BRAFV600E-Positive Melanoma: Participants with melanoma tumors that carried the V600E mutation of the v-raf murine sarcoma viral oncogene homologue B1 (BRAF) received RO5185246 capsules/tablets in MBP formulation at a dose of 960 mg bid until disease progression, death, or withdrawal from the study.
- Extension: BRAFV600E-Positive CRC: Participants with CRC that carried the V600E mutation of the v-raf murine sarcoma viral oncogene homologue B1 (BRAF) received RO5185246 capsules/tablets in MBP formulation at a dose of 960 mg bid until disease progression, death, or withdrawal from the study.
Arm/Group | Dose Escalation: MBP Formulation - 160 mg | Dose Escalation: MBP Formulation - 240 mg | Dose Escalation: MBP Formulation - 320 mg | Dose Escalation: MBP Formulation - 360 mg | Dose Escalation: MBP Formulation - 720 mg | Dose Escalation: MBP Formulation - 1120 mg | Dose Escalation: Original Formulation - 200 mg | Dose Escalation: Original Formulation - 400 mg | Dose Escalation: Original Formulation - 800 mg | Dose Escalation: Original Formulation - 1600 mg | Extension: BRAFV600E-Positive Melanoma | Extension: BRAFV600E-Positive CRC
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 2/3 | 3/5 | 1/7 | 2/6 | 0/6 | 0/6 | 0/10 | 0/4 | 18/32 | 9/21
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/3 | 5/5 | 7/7 | 6/6 | 6/6 | 6/6 | 10/10 | 4/4 | 32/32 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: MBP Formulation - 160 mg (N=4) | Dose Escalation: MBP Formulation - 240 mg (N=4) | Dose Escalation: MBP Formulation - 320 mg (N=3) | Dose Escalation: MBP Formulation - 360 mg (N=5) | Dose Escalation: MBP Formulation - 720 mg (N=7) | Dose Escalation: MBP Formulation - 1120 mg (N=6) | Dose Escalation: Original Formulation - 200 mg (N=6) | Dose Escalation: Original Formulation - 400 mg (N=6) | Dose Escalation: Original Formulation - 800 mg (N=10) | Dose Escalation: Original Formulation - 1600 mg (N=4) | Extension: BRAFV600E-Positive Melanoma (N=32) | Extension: BRAFV600E-Positive CRC (N=21)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 10 | 5
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndroma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: MBP Formulation - 160 mg (N=4) | Dose Escalation: MBP Formulation - 240 mg (N=4) | Dose Escalation: MBP Formulation - 320 mg (N=3) | Dose Escalation: MBP Formulation - 360 mg (N=5) | Dose Escalation: MBP Formulation - 720 mg (N=7) | Dose Escalation: MBP Formulation - 1120 mg (N=6) | Dose Escalation: Original Formulation - 200 mg (N=6) | Dose Escalation: Original Formulation - 400 mg (N=6) | Dose Escalation: Original Formulation - 800 mg (N=10) | Dose Escalation: Original Formulation - 1600 mg (N=4) | Extension: BRAFV600E-Positive Melanoma (N=32) | Extension: BRAFV600E-Positive CRC (N=21)
Fatigue (General disorders) | 1 | 2 | 1 | 4 | 3 | 4 | 2 | 3 | 6 | 0 | 22 | 12
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 9 | 6
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fibrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 6 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3 | 2 | 1 | 2 | 1 | 3 | 2 | 9 | 9
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 6 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 6 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 7 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 13 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 9 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 6
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 1 | 2 | 3 | 0 | 2 | 0 | 0 | 8 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 3 | 2 | 2 | 1 | 1 | 0 | 13 | 5
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 4 | 0 | 6 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 2 | 0 | 1 | 10 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 8 | 3
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 7 | 2
Blood uric acid increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 2 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 5 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 3
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 4 | 0
Xerosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Local Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood Phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Blood Phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Protein Total Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 2 | 3 | 2 | 1 | 2 | 0 | 14 | 7
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 3 | 2 | 1 | 2 | 1 | 2 | 2 | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 11 | 8
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 3 | 1 | 1 | 12 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
faeces pale (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip Swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue atrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
CSF pressure increase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothombin time shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 5 | 4 | 0 | 0 | 2 | 1 | 17 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 1 | 4 | 0 | 0 | 0 | 1 | 18 | 5
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 2 | 2 | 0 | 0 | 1 | 0 | 14 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 3 | 1 | 2 | 0 | 0 | 2 | 0 | 8 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 9 | 5
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 6 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 4 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 10 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 8 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 6 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Campbell de Morgan spots (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 3 | 3 | 1 | 0 | 1 | 0 | 22 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 9 | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Musculoskeletal chest pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 12 | 6
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 4 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 5 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 6 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaethesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 2 | 3 | 1 | 2 | 2 | 1 | 1 | 9 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 7 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 10 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Visual impairment (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Altered visual depth perception (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 4 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mental status change (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 8 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 10 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 10 | 6
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 4 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Deyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal lesion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Trachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 4 | 6
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.